CLINICAL TRIAL: NCT00520286
Title: Phase2, Double-blind, Placebo-controlled Trial of Modafinil for the Treatment of Methamphetamine Dependence
Brief Title: Phase 2, Multi-Center Trial of Modafinil for Methamphetamine Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIDA-CSP-1026-1
Record Dates: First submitted 2007-08-23; First posted 2007-08-24 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-02

CONDITIONS: Methamphetamine Dependence
Keywords: Methamphetamine Dependence
MeSH Terms: interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Modafinil (Active Comparator): Participants will receive a Modafinil 200 mg or 400 mg tablet one time per day for 12 weeks
  Interventions: Drug: Modafinil
- Placebo (Placebo Comparator): Participants will receive a matching Modafinil placebo 200 mg or 400 mg tablet one time per day for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Modafinil — 200 mg or 400 mg /daily
  Arms: Modafinil
Drug: Placebo — Placebo / daily
  Arms: Placebo

SUMMARY:
The purpose of this study will be to examine the safety and efficacy of modafinil in increasing number of methamphetamine non-use weeks in subjects with methamphetamine dependence.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of modafinil in reducing methamphetamine use in subjects with methamphetamine dependence. It is hypothesized that modafinil, compared to placebo, will be associated with an increase in the number of methamphetamine non-use weeks over time as measured by quantitative urine analysis for methamphetamine.

ELIGIBILITY:
Inclusion Criteria:

* Must be between the ages of 18 and 65
* Methamphetamine dependent as defined by DSM-IV criteria
* Must be in good general heath with a history of methamphetamine use at screening
* Must be able to provide written informed consent
* If female and of child bearing potential, must agree to use birth control.

Exclusion Criteria:

* Please contact site for more information

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2007-12; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elkashef, M.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (8):
- United States (8):
  - South Bay Treatment Center, San Diego, California
  - Matrix Institute on Addictions, Tarzana, California
  - Torrance Site, Torrance, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - John A. Burns School of Medicine, Honolulu, Hawaii
  - Powell Chemical Dependency Center, Des Moines, Iowa
  - START Research and Treatment, Kansas City, Missouri
  - Salt Lake City VA Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Anderson AL, Li SH, Biswas K, McSherry F, Holmes T, Iturriaga E, Kahn R, Chiang N, Beresford T, Campbell J, Haning W, Mawhinney J, McCann M, Rawson R, Stock C, Weis D, Yu E, Elkashef AM. Modafinil for the treatment of methamphetamine dependence. Drug Alcohol Depend. 2012 Jan 1;120(1-3):135-41. doi: 10.1016/j.drugalcdep.2011.07.007. Epub 2011 Aug 12. PMID 21840138

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Modafinil | Placebo
Started | 142 | 68
Completed | 76 | 36
Not Completed | 66 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modafinil | Placebo | Total
Number analyzed (Participants) | 142 | 68 | 210
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.6 (17.3) | 39 (8.6) | 39 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 30 | 86
  Male | 86 | 38 | 124
Region of Enrollment [Number; unit: participants]
  United States | 142 | 68 | 210

OUTCOME MEASURES:

1. Primary Outcome: Abstinence (Week 1 - 12)
Description: Number of participant who abstained from methamphetamine from weeks 1 through 12
Time Frame: Weeks 1 - 12
Measure: Count of Participants; unit: Participants
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 142 | 68
Participants
  Week 1 | 27 | 14
  Week 2 | 38 | 13
  Week 3 | 39 | 13
  Week 4 | 46 | 15
  Week 5 | 41 | 16
  Week 6 | 39 | 15
  Week 7 | 34 | 14
  Week 8 | 40 | 16
  Week 9 | 35 | 17
  Week 10 | 34 | 14
  Week 11 | 37 | 16
  Week 12 | 34 | 17

2. Secondary Outcome: Reduction of Craving
Description: Number of subjects with 21 or more consecutive days of abstinence
Time Frame: 21 days
Measure: Count of Participants; unit: Participants
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 142 | 68
Participants | 32 | 10

ADVERSE EVENTS:
Arm/Group | Modafinil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/142 | 5/68
Other Adverse Events (participants affected / at risk) | 128/142 | 54/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modafinil (N=142) | Placebo (N=68)
Leg infection (Infections and infestations) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1)
chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Celluitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Compartment syndrome left forearm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modafinil (N=142) | Placebo (N=68)
Headache (Nervous system disorders) | 60 (175) | 30 (63)
Nausea (Gastrointestinal disorders) | 23 (32) | 8 (13)
Hypertension (Vascular disorders) | 55 (104) | 23 (60)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No